CLINICAL TRIAL: NCT02920047
Title: A Randomized, Open-label, Single Dose, 3x3 Partial Replicated Crossover Study to Evaluate the Pharmacokinetics and Safety/Tolerability Between a Fixed Dose Combination of Fimasartan/Amlodipine and Co-administration of Fimasartan and Amlodipine in Healthy Male Volunteers
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety of Fimasartan and Amlodipine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BR-FAC-CT-102
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence A (Experimental): Period 1(Treatment A) - Period 2(Treatment A) - Period 3(Treatment B)
  There will be a washout of 14 days between the each period.
  Interventions: Drug: Fimasartan/Amlodipine; Drug: Fimasartan + Amlodipine
- Sequence B (Experimental): Period 1(Treatment A) - Period 2(Treatment B) - Period 3(Treatment A)
  There will be a washout of 14 days between the each period.
  Interventions: Drug: Fimasartan/Amlodipine; Drug: Fimasartan + Amlodipine
- Sequency C (Experimental): Period 1(Treatment B) - Period 2(Treatment A) - Period 3(Treatment A)
  There will be a washout of 14 days between the each period.
  Interventions: Drug: Fimasartan/Amlodipine; Drug: Fimasartan + Amlodipine

INTERVENTIONS:
Drug: Fimasartan/Amlodipine — Treatment B
Drug: Fimasartan + Amlodipine — Treatment A

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety when administrated Fimasartan/Amlodipine and when co-administrated Fimasartan and Amlodipine.

DETAILED DESCRIPTION:
This is an open-label, randomized, 3x3 partial replicated crossover study to evaluate the pharmacokinetics and safety/tolerability. Within each period, randomized subjects will be 2 dosing regimens with a fixed dose combination of Fimasartan/Amlodipine and co-administration of Fimasartan and Amlodipine.

ELIGIBILITY:
Inclusion Criteria:

1. Male 19-50 years of age.
2. Body mass index (BMI) ≥ 18 and ≤ 27 kg/m2 at screening.
3. Medically healthy with no clinically significant medical history.
4. Understands the study procedures in the Informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease.
2. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
3. Seated blood pressure is less than 100/65 mmHg or greater than 140/90 mmHg at screening.
4. Plasma donation within a month prior to the first dose of study drug.
5. Participation in another clinical trial within 3 months prior to the first dose of study drug(s).

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cmax and AUClast of Fimasartan, Amlodipine | Time Frame: 0~144 hour after medication

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No